CLINICAL TRIAL: NCT01462968
Title: Interruptions in the Coagulationsystem in Relation With Cardiac Surgery -A Randomized Study Comparing Two Heparinization Strategies During On-pump Cardiac Surgery
Brief Title: Interruptions in the Coagulationsystem in Relation With Cardiac Surgery - A Study Comparing Two Heparinization Strategies During On-pump Cardiac Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never started due to problems with Laboratory facilities in collaborating center
Sponsor: Aalborg University Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jan Jesper Andreasen, Professor, MD, PhD, Professor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N-20110037
Record Dates: First submitted 2011-10-17; First posted 2011-11-01 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2011-10

CONDITIONS: Cardiac Surgery
Keywords: Heparin treatment during cardiac surgery; Heparin reversal after cardiac surgery; Thrombin generation; Endogenous Thrombin potential

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activated clotting time (ACT) group (Active Comparator): heparinization measured as activated clotting time during surgery
  Interventions: Device: Activated clotting time versus blood-heparin concentration
- Hepcon group (Experimental): heparinization measured as heparin concentration in the blood during surgery
  Interventions: Device: Activated clotting time versus blood-heparin concentration

INTERVENTIONS:
Device: Activated clotting time versus blood-heparin concentration — Activated clotting time used for heparinization strategy during cardiag surgery versus blood-heparin concentration
  Other Names: ACT; Hemochron Signature Elite; Hepcon; HMS

SUMMARY:
The purpose of this study is to find the heparinization method, which

1. affect the heparin-protaminsulfate ratio in the best way to achieve haemostasis
2. gives the smallest change in endogenous thrombin potential (ETP)postoperative compared to preoperative (deltaETP) as an indicator for haemostatic activation during cardiac surgery.

The hypothesis is that the deltaETP is larger in the Haemochron Signature Elite group than in the Hepcon-group because of the heparinization-method. Therefore there is a potential higher risk for use of bloodproducts postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Elective on-pump coronary artery bypass grafting (CABG) single procedure
* Elective aortavalve replacement (AVR) (single procedure)

Exclusion Criteria:

* Emergency procedures
* Children and youngsters less than 18 years
* Pregnancy
* Less than 2 days break with platelet inhibiting drugs (acetylsalicylic acid, NSAID, clopidogrel, serotonin reuptake inhibitors)
* Less than 2 days break with AC-treatment (warfarin, heparin, coumarin etc)
* Known coagulopathy
* Endocarditis
* Preoperative anaemia
* Dialysis patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Delta Thrombingeneration | Timeframe is from Start of surgery to 4 hours after end of surgery, average time 9 hours.
  Postoperative versus preoperative thrombingeneration evaluated by Endogenous Thrombin Potential,peak Thrombin level and Lagtime by using a Thromboscope

SECONDARY OUTCOMES:
peroperative heparine/protaminesulphate ratio | The timeframe is from the first heparin is given to the neutralization with protamine sulfate, average time 4 hours
Platelet function | Timeframe is from Start of surgery to 4 hours after end of surgery, average time 9 hours.
  Platelet aggregation measured by Multiplate platelet function analyzer
Thromboelastometry | Timeframe is from Start of surgery to 4 hours after end of surgery, average time 9 hours.
  We are looking at the parameters: Clottingtime, Clot formation time and maximum velocity,maximum clot firmness
Standard coagulationtests | Timeframe is from Start of surgery to 4 hours after end of surgery, average time 9 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne de Neergaard, Perfusionist, Principal Investigator — Heart-Lung surgery unit, Aalborg Hospital, Aarhus University Hospital, Hobrovej 18-22, DK-9000 Aalborg
Locations (1):
- Aalborg Hospital, Aalborg, Aalborg, Denmark